CLINICAL TRIAL: NCT02383537
Title: Biological Changes in the Adipose Tissue (RNA Profile) Among Pregnant Women With Diabetes
Brief Title: Biological Changes in the Adipose Tissue Among Pregnant Women With Diabetes
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Other Study IDs: 0633-14-HMO
Record Dates: First submitted 2015-03-04; First posted 2015-03-09 (Estimated); Last update posted 2016-09-02 (Estimated); Status verified 2015-03

CONDITIONS: Pregnancy; Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Pregnant women with diabetes: Pregnant women with diabetes type 1, type 2 or gestational diabetes
  Interventions: Other: Diabetes
- Healthy pregnant women: Healthy pregnant women with no underlying illness

INTERVENTIONS:
Other: Diabetes — the trial is observational with no intervention
  Groups: Pregnant women with diabetes

SUMMARY:
The aim of the research is to study the effect of miRNA, fat tissue and insulin resistance on the pathophysiology of diabetes during pregnancy. During the study fat tissue, Umbilical cord blood, placenta tissue and subcutaneous fat will be taken from pregnant diabetic woman over going a C-section. Healthy pregnant women will serve as a control group.

DETAILED DESCRIPTION:
The aim of the research is to study the effect of miRNA, fat tissue and insulin resistance on the pathophysiology of diabetes during pregnancy. During the study:

1. fat tissue, Umbilical cord blood, placenta tissue and subcutaneous fat will be taken from pregnant diabetic woman over going a C-section.
2. Bloods will be analyzed for insulin, c-peptide, glucose and fat profile
3. Placenta and fat tissue will be analyzed for miRNA and total RNA
4. Clinical and anthropometric measurements will be taken from the mother
5. Placenta status will be taken

ELIGIBILITY:
Inclusion Criteria:

* age 18-45
* pregnant
* signed consent form
* going through an elective C-section
* Diabetic
* reference group: healthy women with no background illness

Exclusion Criteria:

* <18 or >45
* chronic illness that may effect the outcome
* polypharmacy

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant women with diabetes. Healthy women will serve as a reference group
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2017-04; Primary Completion 2019-02 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
miRNA profiling | samles are taken during C-section samples will be analyzed after completion of collection

CONTACTS AND LOCATIONS:
Overall Officials: Uriel Elchalal, Professor, Principal Investigator — Hadassah Ein Keren; Ram Weiss, Professor, Principal Investigator — Hebrew University